CLINICAL TRIAL: NCT04551456
Title: Randomised, Double-blind, Placebo-controlled, Intravenous Infusion Human Wharton' Jelly-derived Mesenchymal Stem Cells in Patients With Coronary Artery Disease
Brief Title: WJMSCs Anti-inflammatory Therapy in Coronary Artery Disease
Acronym: WANICHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NavyGHB-007
Record Dates: First submitted 2019-12-12; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; anti-inflammatory therapy; human umbilical cord Wharton's jelly-derived MSCs (WJMSCs)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Arms Placebo Comparator: WANICAD Trial are as a 3 arm trial comparing standard of care plus placebo to either standard of care plus WJMSC one or three times infusion with participants allocated to each study arm in a 1:1:1 ratio
Who Masked: Participant, Investigator
Masking Description: Physicians and other clinical personnel remained blind to the treatment assignment throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Infusion PBS (Placebo Comparator): The investigators performed a double-blind, placebocontrolled trial, randomly assigning 100 patients with coronary artery disease to have standard of care plus placebo. Participants allocated to each study arm in a 1:1:1 ratio, to investigate the therapeutic efficacy and safety of WJMSCs in patients with coronary artery disease.
  Assigned Interventions:
  Biological/Vaccine: Biological/Vaccine: WJMSCs Vs.placebo
  Interventions: Biological: Intravenous infusion human umbilical Wharton's jelly-derived mesenchymal stem Cell or placebo PBS
- Single dose Infusion WJMSCs (Experimental): The investigators performed a double-blind, placebocontrolled trial, randomly assigning 100 patients with coronary artery disease to compare standard of care plus placebo to standard of care plus one time or three times in doses of 1x106 /kg of WJMSCs. Participants allocated to each study arm in a 1:1:1 ratio, to investigate the therapeutic efficacy and safety of WJMSCs in patients with coronary artery disease.
  Biological/Vaccine:
  WJMSCs Vs.placebo
  Interventions: Biological: Intravenous infusion human umbilical Wharton's jelly-derived mesenchymal stem Cell or placebo PBS
- Infusion WJMSCs multiple doses (Experimental): The investigators performed a double-blind, placebocontrolled trial, randomly assigning 100 patients with coronary artery disease to compare standard of care plus placebo to one time or three times at 30-day intervals for equal doses of 1x106 /kg of WJMSCs. Participants allocated to each study arm in a 1:1:1 ratio, to investigate the therapeutic efficacy and safety of WJMSCs in patients with coronary artery disease.
  Biological/Vaccine:
  WJMSCs Vs.placebo
  Interventions: Biological: Intravenous infusion human umbilical Wharton's jelly-derived mesenchymal stem Cell or placebo PBS

INTERVENTIONS:
Biological: Intravenous infusion human umbilical Wharton's jelly-derived mesenchymal stem Cell or placebo PBS — Randomised, Double-blind, Placebo-controlled, Intravenous Infusion HumanWharton' Jelly-derived Mesenchymal Stem Cells in Patients With Coronary Artery Disease
  Other Names: Intravenous infusion WJMSCs or placebo

SUMMARY:
As biologic, epidemiologic, and clinical trial data have demonstrated, inflammation is a key driver of atherosclerosis. Recently, a gigantic proof-of-concept trial, CANTOS has demonstrated that inflammation of atherosclerosis can be effectively modulated by Canakinumab. However, fatal infections encountered and high cost in CANTOS. There is, therefore, a clear need for cheaper and safe alternatives. The latest cell biological studies have demonstrated that mesenchymal stem cells have a unique immunomodulatory function. MSCs contribute to a critical role in regulating the inflammatory microenvironment and interacting with immune cells and induce anti- inflammatory macrophages, inhibit foam cell formation, which could reduce atherosclerosis in pre-clinical studies. Therefore, in this randomized, controlled trial, our aim was to assess the safety and the anti-inflammatory efficacy of intravenous infusion human umbilical Wharton's jelly-derived mesenchymal stem Cell (WJMSC) in patients with coronary artery atherosclerosis disease.

DETAILED DESCRIPTION:
As biologic, epidemiologic, and clinical trial data have demonstrated, inflammation is a key driver of coronary artery atherosclerosis, which is associated with pathologic injury and dysregulation of the endothelial cells lining the luminal wall of arteries, accumulation of lipids, macrophages, smooth muscle cells, "foam cells", and aggregated platelets at the arterial luminal wall, resulting in plaque formation. Circulating biomarkers of inflammation, including high-sensitivity C-reactive protein (hsCRP) and interleukin-6 (IL-6), are associated with increased risk of cardiovascular events independent of cholesterol and other traditional risk factors. Recently, a gigantic proof-ofconcept trial CANTOS (Canakinumab Anti-inflammatory Thrombosis Outcomes Study) showed that an antibody that neutralizes IL (interleukin)-1β can reduce recurrent cardiovascular events in secondary prevention, which provides intriguing support for the inflammatory hypothesis of atherosclerosis. Moreover, another agent widely used to treat inflammatory conditions, colchicine,the LoDoCo study (Low-Dose Colchicine) trial has also showed a highly significant reduction in recurrent cardiovascular events over a 3-year follow-up, which also showed promise anti-inflammation in coronary artery disease. Therefore, these studies has demonstrated beyond doubt that inflammation plays a role in the development of atherothrombosis and, more importantly, that it can be effectively modulated.

However, fatal infections encountered and high cost in CANTOS. Colchicine causes gastrointestinal distress sufficient to warrant discontinuation of the medication in over 10% of individuals, the both of which severely limits the wide range of clinical applications. Moreover, more recent clinical evidence from the Cardiovascular Inflammation Reduction Trial (CIRT) has come to challenge the above presented clinical data. low-dose MTX, when compared with placebo, failed to reduce the adverse CV events comprising the original primary end point regarding the cardioprotective effects of MTX. Evidence suggested that the inconsistent cardioprotective effects of different anti-inflammatory agents may be a reflection of the distinct pathways targeted. Atherosclerosis is a chronic inflammatory and immune disease involving multiple cell types, including monocytes, macrophages, T-lymphocytes, endothelial cells, smooth muscle cells and mast cells (MCs). Thus, therapies seek to target the intricate balance between pro- and anti-inflammatory pathways in an attempt to limit inflammation injury.

The latest cell biological studies have demonstrated that mesenchymal stem cells have a unique immunomodulatory function. In low-density lipoproteinreceptor knockout mice atherothrombosis models, MSC-treated mice displayed a signifcant 33% reduction in circulating LY-6C hei monocytes, a 77% reduction of serum CCL2 levels, and signifcantly affected lesion development, which was reduced by 33% in the aortic root. These lesions contained 56% less macrophages and showed a 61% reduction in T cell numbers. MSCs contribute to a critical role in regulating the inflammatory microenvironment and interacting with immune cells, including T cells, B cells, natural killer (NK) cells, and dendritic cells (DCs). MSC induce anti- inflammatory macrophages, inhibit foam cell formation, suppress immune responses of endothelial cells and innate lymphoid cells, and increase phagocytic capacity, which indirectly suppresses T cell proliferation. More recently, the paracrine potency might vary with sources and microenvironment of MSCs. MSCs isolated from fetal tissues such as umbilical cord (UC) and UC-blood (UCB) were shown to have increased secretion of anti-inflammatory factors (TGF-β,IL-10) and growth factors than MSCs obtained from adult adipose tissue or bone marrow. Our previous research found that the expression characteristics of special immunomodulatory genes of human umbilical cord Wharton's jelly-derived MSCs (WJMSCs) .We found WJMSCs transplantation significantly reduced the number of inflammatory macrophages (M1), increased the number of anti-inflammatory macrophages (M2) and prevented the expansion of AMI during early stage of AMI in mouse AMI models. At present, many studies have demonstrated WJMSC possess a robust immunomodulatory potential and anti-inflammatory effects through release of secretome consisting of a diverse range of cytokines, chemokines, and extracellular vesicles (EVs), the cross talk and interplay of WJMSCs and local environment reversely control and regulate the paracrine activity of MSCs. Thus WJMSCs are important regulators of immune responses and may hold great potential to be used as a therapeutic in atherosclerosis. In particular safety and feasibility of WJMSCs transplant have been clearly proved by us and other studies.

Given the current evidence, systemic paracrinemediated anti-inflammatory effects of WJMSCs can drive beneficial in therapy of atherosclerosis. These concepts lead to a potentially transformative strategy that intravenous delivery of WJMSCs, through systemic anti-inflammatory mechanisms.Therefore, the investigators performed a double-blind, placebo- controlled trial, randomly assigning 300 patients with coronary artery disease to receive three times at 30-day intervals for equal doses of 1x106 /kg of WJMSCs or placebo , to investigate the therapeutic efficacy and safety of WJMSCs in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at Visit 1;
2. Patient must provide written informed consent;
3. Have a diagnosis of coronary artery atherosclerotic disease as defined by any of the following 3 criteria:

   1. Previous MI is documented by a clinical history or documented either by hospital records or by evidence that includes an elevation of cardiac enzymes and/or electrocardiogram (ECG) changes consistent with MI.
   2. All patients underwent invasive coronary angiography at the time of presentation and were revascularized if clinically indicated, or these patients underwent coronary CTA
   3. Multivessel coronary disease confirmed by coronary angiography or CTA

Exclusion Criteria:

1. Evidence of a life-threatening arrhythmia (ventricular tachycardia or complete heart block) on screening ECG..
2. Have a hematologic abnormality as evidenced by hematocrit <25% , white blood cell <2500/u L or platelet values<100000/u L without another explanation.
3. Have liver dysfunction, as evidenced by enzymes (aspartate aminotransferase and alanine aminotransferase) >3× the upper limits of normal.
4. Have a coagulopathy (international normalized ratio>1.3) not because of a reversible cause (ie, coumadin).
5. Be an organ transplant recipient.
6. Have a clinical history of malignancy within 5 y except curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
7. Have a noncardiac condition that limits lifespan to <1y.
8. Have a history of drug or alcohol abuse within the past 24 m.
9. Be serum positive for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C.
10. Be a female who is pregnant, nursing, or of childbearing potential who is not practicing effective contraceptive methods.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary end point was checking incidence of adverse events (AEs) within 12 months, | up to 12 months
  Including death from any cause; a composite of major adverse cardiovascular events of nonfatal myocardial infarction, nonfatal stroke, or cardiovascular death and hospitalization for unstable angina that led to urgent coronary revascularization;

SECONDARY OUTCOMES:
The secondary end point was measuring low attenuation plaque volume LAPV | up to 10 months
  The secondary end point was efficacy, which was assessed in terms of the change in low attenuation plaque volume LAPV by Coronary computed tomography angiography (coronary CTA) from baseline to 12 months.
The secondary end point was efficacy 2 | up to 10 months
  The level of high-sensitivity C-reactive protein (hsCRP) from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Ru Gao, MD, Study Chair — Navy General Hospital, Beijing